CLINICAL TRIAL: NCT02704507
Title: Addition of a Topical Steroid to a Topical Retinoid: a Randomized, Split-face, Placebo-controlled, Double-blind, Single-center Clinical Study
Brief Title: Addition of a Topical Steroid to a Topical Retinoid in Acne Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Michael Kolodney, Section Chief Dermatology, Carilion Clinic Dermatology, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1771
Record Dates: First submitted 2016-02-13; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Acne
Keywords: tretinoin; topical steroid; irritation; retinoid induced irritation
MeSH Terms: conditions — Acne Vulgaris | interventions — Triamcinolone; Tretinoin; Emollients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Topical steroid (Experimental): Topical retinoid plus topical steroid applied daily to half of the face for 4 weeks, followed by 4 weeks of topical tretinoin. Patients will be randomized to which side receives the topical steroid.
  Interventions: Drug: Triamcinolone; Drug: Tretinoin
- Topical emollient (Placebo Comparator): Topical retinoid plus topical emollient applied daily to the opposite half of the face for 4 weeks, followed by 4 weeks of topical tretinoin.
  Interventions: Drug: Tretinoin; Drug: Emollient

INTERVENTIONS:
Drug: Triamcinolone — topical application nightly to half the face for 4 weeks
  Arms: Topical steroid
Drug: Tretinoin — topical application nightly for 8 weeks
Drug: Emollient — topical application nightly to half the face for 4 weeks
  Arms: Topical emollient

SUMMARY:
A randomized, split-face, placebo-controlled, double-blind, single-center clinical trial comparing topical retinoid on half the face and retinoid plus topical steroid on the other half.

DETAILED DESCRIPTION:
A randomized, split-face, placebo-controlled, double-blind, single-center clinical trial wherein 20 patients received daily 0.05% tretinoin with one half of the face receiving triamcinolone 0.025% and the other half an inert emollient for 4 weeks. Subjects continued applying tretinoin 0.05% daily to the bilateral face without triamcinolone or emollient for an additional 4 weeks. Investigator's Global Assessment, lesion counts, and study subject's self-assessments of burning/stinging, itching, erythema, and dryness/scaling will be collected at 1, 2, 4, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin types I, II, or III
* Will and ability to discontinue use of topical medicines on the face for study duration
* Capability to understand and provide informed consent

Exclusion Criteria:

* Use of oral retinoids within previous 6 months
* Use of corticosteroids on the face or systemic corticosteroids within previous 4 weeks
* Any additional facial skin condition (i.e., rosacea, seborrheic dermatitis, etc.)
* Female participants who are pregnant, nursing, or planning pregnancy while participating in the study
* Hypersensitivity to ingredients in study formulations
* Existence of an underlying condition that an investigator feels would hinder a participant's ability to complete the study or appropriately follow directions

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in subject-assessed itching and burning/stinging assessed by a 0-3 score over 8 weeks | baseline, weeks 1,2, 4, and 8
  Subject will given a questionnaire to assess itching and burning/stinging on each side of the face on a 0-3 scale: (0) None- Normal, no discomfort; (1) Slight- A noticeable discomfort that causes intermittent awareness; (2) Moderate- A noticeable discomfort that causes intermittent awareness and interferes occasionally with normal daily activities; (3) Strong- A definite continuous discomfort that interferes with normal daily activities.
Change in physician-assessed erythema scores assessed by a 0-4 scale over 8 weeks. | baseline, weeks 1,2, 4, and 8
  Physicians will assess each side of subjects' face for erythema: (0) absent: no redness; (1) slight: Faint red or pink coloration, barely perceptible; (2) mild: light red or pink coloration; (3) moderate: medium red coloration; (4) severe: beet red coloration.
Change in physician-assessed dryness scores assessed by a 0-4 scale over 8 weeks. | baseline, weeks 1,2, 4, and 8
  Physicians will assess each side of subjects' face for dryness: (0) absent: none; (1) slight: barely perceptible dryness with no flakes or fissure formation; (2) mild: easily perceptible dryness with no flakes or fissure formation; (3) moderate: easily noted dryness and flakes but no fissure formation; (4) severe:easily noted dryness with flakes and fissure formation.
Change in physician-assessed peeling scores assessed by a 0-4 scale over 8 weeks. | baseline, weeks 1,2, 4, and 8
  Physicians will assess each side of subjects' face for peeling: (0) absent: no peeling; (1) slight:mild localized peeling; (2) mild: mild and diffuse peeling; (3) moderate: moderate and diffuse peeling; (4) severe:moderate to prominent, dense peeling.

SECONDARY OUTCOMES:
Change in physician-assessed inflammatory and non-inflammatory lesion counts over 8 weeks | baseline, weeks 1,2, 4, and 8
  Physicians will count the inflammatory and non-inflammatory lesions on each side of the face over 8 weeks.
Change in physician-assessed global acne scores over 8 weeks. | baseline, weeks 1,2, 4, and 8
  Physicians will grade each side of the subject's face on the "Global Acne Score" 0-5 over 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kolodney, MD, PhD, Principal Investigator — Carilion Clinic